CLINICAL TRIAL: NCT00011453
Title: NQO1 in Protection Against Benzene Toxicity
Brief Title: Protection Against Benzene Toxicity
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9554-CP-001
Record Dates: First submitted 2001-02-21; First posted 2001-02-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Leukemia; Aplastic Anemia
Keywords: NQO1; DT-diaphorase; Benzene; Leukemia; Aplastic anemia
MeSH Terms: conditions — Leukemia; Anemia, Aplastic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
We are investigating the role of an enzyme (NQO1) in protection against the bone marrow toxicity of the occupational and environmental toxicant benzene. All of the proposed studies involve use of human bone marrow cells in-vitro to define mechanisms of NQO1-mediated protection. Cells are obtained from healthy volunteers and protocols have undergone IRB review and approval.

ELIGIBILITY:
Healthy adult volunteers with blood counts in normal ranges and without evidence of hepatitis or HIV infection.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States